CLINICAL TRIAL: NCT07294599
Title: Morning Versus Evening Patching in Childhood Amblyopia-A Randomized Clinical Trial
Brief Title: Morning Versus Evening Patching in Childhood Amblyopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yarmouk University (Other)
Responsible Party: Principal Investigator, Rami Alomari, Associate professor, Yarmouk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB/2025/318
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Amblyopia
Keywords: Morning patching; Evening patching; Amblyopia; Clinical trial; Anisometriopia; Strabismus
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Intervention Model Description: Intervention model: Parallel-group, randomized assignment. Children with unilateral amblyopia will be randomized 1:1 to one of two arms: (1) morning patching (08:00-10:00 daily) or (2) evening patching (17:00-19:00 daily). Participants remain in their assigned arm for the full 6-month study and receive 2 hours/day occlusion with near-vision tasks. Outcomes (visual acuity ± stereoacuity) are assessed at baseline, 3 months (midpoint), and 6 months (final). Stratified randomization (by age group 4-<6 vs 6-8 years, baseline VA severity, and amblyopia type) ensures balanced prognostic variables across arms. The purpose is efficacy comparison - to determine whether timing of daily occlusion (morning vs evening) affects improvement in the amblyopic eye after 6 months.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments (visual acuity, stereoacuity, ocular alignment) will be performed by trained examiners (e.g., optometrists/orthoptists) who are not involved in randomization, patching-instructions, or adherence monitoring, and who will remain masked to the child's assignment (morning vs evening patching). Allocation will be concealed via a central computer-generated randomization list; the enrolling investigator will not communicate assignment to the assessor. Standard operating procedures (chart, lighting, refractive correction, instructions) will be used uniformly. Data entered in the database will use non-descriptive group codes ("Group A" / "Group B"), and the statistician will remain blinded until the database is locked and primary analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning patching (Experimental): Daily occlusion: 2 hours/day between 08:00-10:00.
  During patching: child performs near-vision activities (e.g. reading, puzzles, coloring).
  Duration: 6 months (unless withdrawal criteria met).
  Interventions: Behavioral: eye-patching
- Evening patching (Experimental): Daily occlusion: 2 hours/day between 17:00-19:00.
  During patching: same near-vision tasks as Arm 1.
  Duration: 6 months (unless withdrawal criteria met).
  Interventions: Behavioral: eye-patching

INTERVENTIONS:
Behavioral: eye-patching — is a non-invasive treatment for Amblyopia ("lazy eye") in children. It involves covering (patching) the stronger, "good" eye so that the weaker (amblyopic) eye is forced to work. This encourages the brain to rely on the amblyopic eye, helping to strengthen its visual pathways.
  Other Names: occlusion therapy

SUMMARY:
To determine whether the time of day at which daily occlusion (patching) is administered - morning (08:00-10:00) versus evening (17:00-19:00) - affects the amount of visual-acuity improvement in the amblyopic eye in children with unilateral amblyopia.

Rationale:

While occlusion therapy remains the mainstay for treatment of childhood amblyopia, existing trials have focused on patching duration, not on the timing of occlusion. Diurnal or chronobiological factors - such as fluctuations in neuroplasticity, attention, compliance, or visual demand during the day - may influence the efficacy of patching. Understanding whether timing matters could help optimize occlusion therapy, improve outcomes, and reduce treatment burden.

DETAILED DESCRIPTION:
Study Type: Prospective, randomized, parallel-group clinical trial.

Participants: Children aged 4-8 years with unilateral amblyopia; amblyopic-eye BCVA between 0.17-0.67 decimal (≈ 6/36-6/9); fellow-eye BCVA ≥ 0.80 decimal; refractive-dominant or strabismic/mixed amblyopia. Parental/guardian consent required.

Randomization & Stratification: Participants randomized 1:1 to "Morning patching" vs "Evening patching" arms. Stratified by age (4-<6 vs >=6-8), baseline visual acuity or amblyopia severity (moderate 6/36-<6/12 vs mild 6/12-6/9), and amblyopia type (refractive-dominant vs strabismic/mixed) - to ensure balance across key prognostic variables.

Intervention: Daily occlusion of the non-amblyopic eye for 2 continuous hours, at assigned time window (Morning: 08:00-10:00; Evening: 17:00-19:00). During patching, child engages in near-vision tasks (reading, puzzles, coloring) for 20-30 min or more. Adherence monitored via parent diary/photos. Spectacle correction (if prescribed) maintained throughout.

Follow-up / Assessments:

Baseline exam (BCVA both eyes, refraction, ocular alignment/strabismus assessment, anterior and posterior segment exam, stereoacuity, instructions on patching/adherence, randomization).

Midpoint follow-up at 3 months (BCVA, adherence, adverse events. Telehealth acceptable if in-person not possible.).

Final follow-up at 6 months (BCVA (primary endpoint), stereoacuity, ocular alignment/strabismus assessment, anterior segment exam, adherence data review, adverse events, patching compliance summary.).

Primary Outcome: Change in best-corrected visual acuity (BCVA) of the amblyopic eye from baseline to month 6.

Secondary Outcomes: Stereoacuity improvement, adherence rate (% of days/patching sessions completed).

Statistical Approach: Analysis of covariance (ANCOVA) comparing mean change in BCVA between arms, adjusting for baseline VA and stratification factors. Subgroup analyses by amblyopia type, baseline severity, age group.

Sample Size / Power (Summary):

Target total enrollment ~100 children (≈ 50 per arm), to provide sufficient power to detect a clinically meaningful difference (≈ 1 line difference in BCVA) between morning and evening patching, while allowing for variability, drop-outs, and stratified analyses.

Duration & Timeline:

Each participant will be followed for 6 months of daily patching. The total study duration (from first enrollment to last follow-up) will depend on recruitment rate; estimated duration ~ 7-9 months including recruitment, follow-up, data cleaning, and analysis.

Significance & Expected Impact:

If timing of occlusion influences visual outcome, this could refine occlusion therapy recommendations - potentially improving efficacy, adherence, and convenience for patients and families. The trial may identify a more effective or practical patching schedule, thereby contributing to evidence-based amblyopia management.

ELIGIBILITY:
Inclusion Criteria:

* Age: 4-8 years.
* Unilateral amblyopia.
* Amblyopic-eye BCVA decimal 0.17-0.67 (≈ 6/36-6/9).
* Fellow-eye BCVA ≥ 0.80 decimal (≈ 6/7.5 or better).
* Amblyopia type: refractive-dominant or strabismic/mixed.
* Parent/guardian consent obtained.

Exclusion Criteria:

* Bilateral amblyopia.
* Sensory-deprivation amblyopia (e.g., due to congenital cataract, ptosis, corneal opacity).
* Ocular surgery within the past 6 months, or planned surgery during study.
* Likely poor adherence (e.g., due to social, logistic, or family constraints).

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-12-14 (Estimated); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) of the amblyopic eye | 6 month
  Change in best-corrected visual acuity (BCVA) of the amblyopic eye from baseline to month 6, measured using a standardized logMAR (crowded) chart under full refractive correction, by a masked examiner.

SECONDARY OUTCOMES:
stereoacuity | 6 month
  Change in stereoacuity (arc-seconds unit) from baseline to Month 6 in amblyopic eye in the trial measured using the Titmus Fly Test